CLINICAL TRIAL: NCT03643887
Title: A Phase II Randomized, Double-blind Placebo-controlled Trial of Fecal Microbiota Transplantation for Vancomycin-resistant Enterococcus and Carbapenem-resistant Enterobacteriaceae
Brief Title: Phase II Trial of Fecal Microbiota Transplant (FMT) for VRE and CRE Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding obtained
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: W81XWH18PRMPCTA
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2020-06

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FMT Capsule DE (Experimental): FMT Capsule DE
  Interventions: Drug: FMT Capsule DE
- Placebo Oral Capsule (Placebo Comparator): Placebo Capsule
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: FMT Capsule DE — 30 capsule one-time oral dose
  Arms: FMT Capsule DE
Drug: Placebo oral capsule — 30 capsule one-time oral dose
  Other Names: Placebo
  Arms: Placebo Oral Capsule

SUMMARY:
Vancomycin-resistant Enterococcus (VRE) and carbapenem-resistant Enterobacteriaceae (CRE) are multi-drug resistant organisms (MDROs) associated with healthcare settings and are a high priority for containment in public health. Healthcare-associated infections (HAIs) like VRE and CRE lengthen the duration of a hospital stay, increase the cost of hospitalization, and increase mortality. Because colonization precedes infection, prevention or treatment of VRE/CRE colonization is essential. We propose a treatment approach to promote gut decolonization by VRE and CRE without using antibiotics. Participants enrolled in this study will be randomized a one-time dose of either study drug or placebo, will be followed for 6 months, and will submit stool samples for analysis of several outcomes for the trial.

DETAILED DESCRIPTION:
This is a phase II, double-blind, randomized, placebo controlled trial assessing the effects of one-time oral FMT on the composition and function of the gut microbiome compared to placebo in a population of patients with baseline CRE or VRE gut colonization. Participants will be adults who have had two consecutive positive stool cultures for VRE or CRE and meet all inclusion/exclusion criteria. Patients (N=90) will be randomized at a 1:1 ratio. Randomization will be double-blinded. Each subject will be followed for 6 months. Stool samples will be taken at baseline and from subjects weekly for 4 weeks, then every 4 weeks for 8 weeks, then at 6 months regardless of treatment group. All patients will be asked to complete a stool diary

ELIGIBILITY:
Inclusion Criteria:

* Cognitively intact and willing to provide informed consent
* Willing and able to comply with all study procedures for the duration of the study
* Age 18 years or older
* Two positive stool cultures for CRE or VRE (positive for the same organism on both cultures). The most recent stool culture must be within 14 days of randomization.
* Women of childbearing potential in a sexual relationship with men must use an acceptable method of contraception (including, but not limited to, barrier with additional spermicidal foam or jelly, intrauterine device, hormonal contraception started at least 30 days before enrollment into the study, or intercourse with men who underwent a vasectomy) for 4 weeks following completion of the study treatment.
* Males must agree to avoid impregnation of women during and for 4 weeks following completion of the study treatment through the use of an acceptable method of contraception (including but not limited to, barrier with additional spermicidal foam or jelly or vasectomy).
* Able to take the test capsule successfully with no signs or symptoms of dysphagia.

Exclusion Criteria:

* Admitted to an intensive care unit (ICU) for medical reasons (not just boarding).

Patients residing in a nursing home, long-term care facility or rehabilitation center may be enrolled.

* Patient received antibiotics in the last 48 hours. Patients will be eligible to enroll if antibiotic therapy is discontinued for at minimum 48 hours prior to randomization. Does not include antibiotics used for prophylaxis or topical antibiotics.
* Requires continued antibiotic use or anticipates antibiotic use in the upcoming 4 weeks.
* Unwilling to withhold probiotics for a minimum of 48 hours prior to providing a screening stool sample.
* Previous FMT or microbiome-based products in the last 90 days.
* Active antibiotic-resistant bacteria (ARB) or gastrointestinal infection at time of enrollment.
* Any other gastrointestinal illness including diarrhea.
* Known or suspected toxic megacolon and or known small bowel ileus.
* Bowel obstruction or other gut motility issues as noted by the patient or in the electronic medical record.
* Major gastrointestinal surgery (e.g. significant bowel resection) within 3 months before enrollment not including appendectomy or cholecystectomy.
* History of total colectomy or bariatric surgery.
* Concurrent intensive induction chemotherapy, radiation therapy, or biologic treatment for an active malignancy. Patients on maintenance chemotherapy may be enrolled after consultation with the medical monitor.
* Patients with severe anaphylactic or anaphylactoid food allergy.
* Solid organ transplant recipients ≤90 days post-transplant or on active treatment for rejection.
* Neutropenia (≤500 neutrophils/mL) or other severe immunosuppression. Anti-tumor necrosis factor (anti-TNF) will be permitted. Participants taking glucocorticoids, antimetabolites (azathioprine, 6-mercaptopurine, methotrexate), calcineurin inhibitors (tacrolimus, cyclosporine) and mycophenolate mofetil may be enrolled only after consultation with the medical monitor.
* If At risk of CMV/EBV associated disease (at discretion of investigators, e.g. immunocompromised participant), negative Immunoglobulin G (IgG) testing for cytomegalovirus (CMV) or Epstein Barr Virus (EBV).
* Cognitive impairment at the time of enrollment.
* Expected life expectancy <6 months.
* Inability (e.g. dysphagia) to or unwilling to swallow capsules.
* Unable or unwilling to comply with protocol requirements.
* Any condition that would jeopardize the safety or rights of the patient, would make it unlikely for the patient to complete the study, or would confound the results of the study.
* Females who are pregnant, lactating, or planning to become pregnant during the study.

Female patients of childbearing potential will take a pregnancy test and be excluded if pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Compare incidence of VRE/CRE decolonization between FMT Capsule double encapsuled (DE) and placebo | 6 months
  VRE/CRE decolonization is defined by absence of VRE/CRE on stool culture using standard laboratory techniques.

SECONDARY OUTCOMES:
VRE/CRE infection at Day 3, Day 10, and Week 4 following randomization. | 1 month
  VRE/CRE infection will be defined as an associated bacteremia, urinary tract infection, or would-related infection.
Microbial engraftment assessed by microbial disruption index (MDI) at Day 3, Day 10, and Week 4 following randomization | 1 month
  VRE/CRE type and strain level engraftment, using whole genome sequencing laboratory techniques
Antibiotic resistant bacteria (ARB) decolonization at Day 10 after randomization. | 10 days
  ARB testing will be done with Acuitas (OpGen) MDRO test or a similar platform
Antibiotic resistant bacteria (ARB) infection at Day 3, Day 10, Week 4 after randomization, and time to infection if ARB infection occurs | 1 month
  ARB infection will be defined as extended spectrum beta lactamase clinical infection.
Adverse events/serious adverse events through Day 10, Week 4, and Month 6 following randomization. | 6 months
  Safety of FMT Capsule DE compared to placebo. Incidence of newly acquired transmissible infectious diseases that are considered adverse events of special interest (AESI).

CONTACTS AND LOCATIONS:
Overall Officials: Nasia Safdar, MD PhD, Principal Investigator — Infectious Disease, School of Medicine & Public Health, University of Wisconsin-Madison

IPD SHARING:
Plan to Share IPD: No